CLINICAL TRIAL: NCT00596284
Title: Cognitive Behavior Therapy for Anxiety in Dementia
Brief Title: Cognitive Behavior Therapy for Treating Anxiety in People With Dementia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Melinda Stanley, Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R34MH078925 (NIH); R34MH078925 (NIH); DATR A4-GPS
Record Dates: First submitted 2008-01-04; First posted 2008-01-16 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Anxiety Disorders; Dementia
Keywords: Cognitive Behavior Therapy; Alzheimer's Disease
MeSH Terms: conditions — Anxiety Disorders; Dementia; Alzheimer Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CBT-AD (Experimental): Participants will receive Cognitive Behavioral Therapy of Anxiety in Dementia (CBT-AD)
  Interventions: Behavioral: Cognitive Behavioral Therapy of Anxiety in Dementia (CBT-AD)
- EUC (Active Comparator): EUC will consist of regular ongoing care from healthcare providers and phone assessments at 1-month and 2-month. Following the 6 month assessment, participants in EUC will be offered a half-day Cognitive Behavior Workshop.
  Interventions: Behavioral: Enhanced Usual Care (EUC)

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy of Anxiety in Dementia (CBT-AD) — Cognitive behavioral therapy (CBT) will consist of 8 to 10 sessions over a period of 10 to 12 weeks. Each CBT session will last about 1 hour and will include meeting with a study staff member to discuss anxiety and how to cope with it. Participants will also complete practice activities at home for about 20 minutes per day.
  Arms: CBT-AD
Behavioral: Enhanced Usual Care (EUC) — Following in-person meetings, participants will receive weekly phone calls for 3 months, followed by biweekly phone calls for the next 3 months.
  Arms: EUC

SUMMARY:
This study will evaluate the effectiveness of cognitive behavioral therapy in treating anxiety in older adults with dementia.

DETAILED DESCRIPTION:
Dementia is an illness that causes memory problems; changes in behavior; and difficulty with thinking, making decisions, and carrying out daily activities. Many people with dementia also have anxiety, and yet very little is known about effective treatment strategies for anxiety in this population. Cognitive behavioral therapy (CBT) is a type of psychotherapy that is commonly used to treat anxiety. CBT involves teaching patients skills to help them manage their anxiety, such as relaxation, changing their thoughts, and problem-solving. This study will evaluate the effectiveness of CBT in treating anxiety in older adults with dementia. In addition, the study will determine the effect of the treatment on patients' families and friends, and how families and friends may be able to help patients manage their anxiety. All study participants will name a family member or friend who will also participate in the study.

All participants in this study will answer a preliminary set of questions about anxiety and memory and will then complete a number of activities that involve learning and memory. These evaluations will take approximately 45 minutes. Participants who are selected to continue in the study will answer a second set of questions about mood, memory, concentration, and how they are doing in certain areas of life. These interview questions will take place during 2 sessions and will last a total of approximately 3 hours. Participants will then be randomly assigned to receive either enhanced usual care (EUC) or 8 to 10 sessions of CBT over a period of 10 to 12 weeks. Each CBT session will last about 1 hour and will include meeting with a study staff member to discuss anxiety and how to cope with it. Participants will also complete practice activities at home for about 20 minutes per day. EUC will consist of regular ongoing care from healthcare providers and phone assessments at 1-month and 2-month. Following the 6 month assessment, participants in EUC will be offered a Cognitive Behavior Workshop. Following in-person meetings, CBT participants will receive weekly phone calls for 3 months, followed by biweekly phone calls for the next 3 months. Some of the pretreatment questions will be asked again at 3 months and again 6 months after baseline.

ELIGIBILITY:
Inclusion Criteria:

* Alzheimer's disease that is in the mild or moderate range according to a score of 0.5 to 2.0 on the Clinical Dementia Rating (CDR) Scale
* Significant anxiety as defined by a score of 4 on the Neuropsychiatric Inventory (NPI)
* Agrees to permit participation of a collateral
* English-speaking

Exclusion Criteria:

* Suicidal intent
* Current psychosis or bipolar disorder
* History of substance abuse within 1 month prior to study entry

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2008-01; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Rating Anxiety in Dementia (RAID) and Neuropsychiatric Inventory (NPI)- Anxiety subscales | Measured at pre-treatment, post-treatment, and 3-month follow-up

SECONDARY OUTCOMES:
Quality of Life in Alzheimer's Disease (QOL-AD) | Measured at pre-treatment, post-treatment, and 3-month follow-up
Geriatric Depression Scale (GDS) | Measured at pre-treatment, post-treatment, and 3-month follow-up
Penn State Worry Questionnaire (PSWQ) | Measured at pre-treatment, post-treatment, and 3-month follow-up
Geriatric Anxiety Inventory (GAI) | Measured at pre-treatment, post-treatment, and 3-month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Melinda A. Stanley, PhD, Principal Investigator — Baylor College of Medicine; Jessica Calleo, PhD, Study Director — Baylor College of Medicine
Locations (2):
- United States (2):
  - Baylor College of Medicine, Houston, Texas
  - Michael E. DeBakey Veterans Affairs Medical Center, Houston, Texas